CLINICAL TRIAL: NCT02341638
Title: Randomized, Double-Blinded, Placebo-Controlled Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986141 in Healthy Subjects
Brief Title: Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986141 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CV006-003
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2015-09

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — BMS-986141; Aspirin; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (17):
- Part A Panel 1: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part A Panel 2: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part A Panel 3: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part A Panel 4: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part A Panel 5: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part A Panel 6: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part A Panel 7: BMS-986141 (Experimental): Single dose by mouth as specified
  Interventions: Drug: BMS-986141
- Part A Panel 8: BMS-986141 (Experimental): Single dose by mouth as specified
  Interventions: Drug: BMS-986141
- Part B Panel 1: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part B Panel 2: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part B Panel 3: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part C Panel 1: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part C Panel 2: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part C Panel 3: BMS-986141 or Placebo (Experimental): BMS-986141 or Placebo by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Placebo
- Part D Panel 1: BMS-986141 and Aspirin (Experimental): BMS-986141 and Aspirin by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Aspirin
- Part D Panel 1: Placebo matching BMS-986141 and Aspirin (Placebo Comparator): BMS-986141 placebo and Aspirin by mouth as specified
  Interventions: Drug: Placebo; Drug: Aspirin
- Part E Panel 1: BMS-986141 and Itraconazole (Experimental): BMS-986141 and Itraconazole by mouth as specified
  Interventions: Drug: BMS-986141; Drug: Itraconazole

INTERVENTIONS:
Drug: BMS-986141
  Arms: Part A Panel 1: BMS-986141 or Placebo; Part A Panel 2: BMS-986141 or Placebo; Part A Panel 3: BMS-986141 or Placebo; Part A Panel 4: BMS-986141 or Placebo; Part A Panel 5: BMS-986141 or Placebo; Part A Panel 6: BMS-986141 or Placebo; Part A Panel 7: BMS-986141; Part A Panel 8: BMS-986141; Part B Panel 1: BMS-986141 or Placebo; Part B Panel 2: BMS-986141 or Placebo; Part B Panel 3: BMS-986141 or Placebo; Part C Panel 1: BMS-986141 or Placebo; Part C Panel 2: BMS-986141 or Placebo; Part C Panel 3: BMS-986141 or Placebo; Part D Panel 1: BMS-986141 and Aspirin; Part E Panel 1: BMS-986141 and Itraconazole
Drug: Placebo
  Arms: Part A Panel 1: BMS-986141 or Placebo; Part A Panel 2: BMS-986141 or Placebo; Part A Panel 3: BMS-986141 or Placebo; Part A Panel 4: BMS-986141 or Placebo; Part A Panel 5: BMS-986141 or Placebo; Part A Panel 6: BMS-986141 or Placebo; Part B Panel 1: BMS-986141 or Placebo; Part B Panel 2: BMS-986141 or Placebo; Part B Panel 3: BMS-986141 or Placebo; Part C Panel 1: BMS-986141 or Placebo; Part C Panel 2: BMS-986141 or Placebo; Part C Panel 3: BMS-986141 or Placebo; Part D Panel 1: Placebo matching BMS-986141 and Aspirin
Drug: Aspirin
  Arms: Part D Panel 1: BMS-986141 and Aspirin; Part D Panel 1: Placebo matching BMS-986141 and Aspirin
Drug: Itraconazole
  Arms: Part E Panel 1: BMS-986141 and Itraconazole

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of a single and multiple oral doses of BMS-986141 in healthy subjects.

DETAILED DESCRIPTION:
Maximum Age:

Part A SAD 65 years

Part B MAD 75 years

Part C MAD Japanese 75 years

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. Healthy male and female subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
2. Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI=Weight (kg)/[height(m)]2
3. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and men, ages 18 to 75, inclusive

Exclusion Criteria:

1. Concurrent or use within 2 weeks of study drug administration, of marketed or investigational, drugs as specified in protocol
2. Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Up to 30 days post discontinuation of dosing or last participation in the study
  Serious adverse event (SAE)
  Adverse event (AE)
  Electrocardiogram (ECG)
Tolerability measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Up to 30 days post discontinuation of dosing or last participation in the study
Safety measured by percent of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Up to 30 days post discontinuation of dosing or last participation in the study
Tolerability measured by percent of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Up to 30 days post discontinuation of dosing or last participation in the study

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
Time of maximum observed plasma concentration (Tmax) of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
Concentration at 24 hours (C24) of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
Half-life (T-HALF) of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
AUC accumulation index (AI_AUC) of BMS-986141, BMT-162853, BMT-162856, and BMT-181551; ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose | Up to Day 14
Effective elimination half-life that explains the degree of AUC accumulation observed (T-HALFeff_AUC) of BMS-986141, BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
MR_Cmax of BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
  Ratio of metabolite Cmax to parent Cmax, corrected for molecular weight (MR_Cmax)
MR_AUC(INF) of BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
  Ratio of metabolite AUC(INF) to parent AUC(INF), corrected for molecular weight [MR_AUC(INF)]
MR_AUC(0-T) of BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
  Ratio of metabolite AUC(0-T) to parent AUC(0-T), corrected for molecular weight [MR_AUC(0-T)]
MR_AUC(TAU) of BMT-162853, BMT-162856, and BMT-181551 | Up to Day 14
  Ratio of metabolite AUC(TAU) to parent AUC(TAU), corrected for molecular weight [MR_AUC(TAU)]
Safety of multiple doses of BMS-986141 and aspirin in healthy subjects | Up to 30 days post discontinuation of dosing or last participation in the study
  Safety measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations.
Tolerability of multiple doses of BMS-986141 and aspirin in healthy subjects | Up to 30 days post discontinuation of dosing or last participation in the study
  Tolerability measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations
Safety of BMS-986141 and itraconazole in healthy subjects | Up to 30 days post discontinuation of dosing or last participation in the study
  Safety measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations
Tolerability of BMS-986141 and itraconazole in healthy subjects | Up to 30 days post discontinuation of dosing or last participation in the study
  Tolerability measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - West Coast Clinical Trials, Llc, Cypress, California
  - Ppd Development, Lp, Austin, Texas

REFERENCES:
- [Derived] Merali S, Wang Z, Frost C, Meadows-Shropshire S, Hawthorne D, Yang J, Seiffert D. First-in-human study to assess the safety, pharmacokinetics, and pharmacodynamics of BMS-986141, a novel, reversible, small-molecule, PAR4 agonist in non-Japanese and Japanese healthy participants. Platelets. 2023 Dec;34(1):2222846. doi: 10.1080/09537104.2023.2222846. PMID 37394920
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx